CLINICAL TRIAL: NCT06501222
Title: The Renal Protective Effects of Remote Ischemic Preconditioning in Patients With Chronic Kidney Disease: Randomized, Parallel-controlled, proof-of Concept Trial
Brief Title: The Renal Protective Effects of Remote Ischemic Preconditioning in Patients With Chronic Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuanjun Yang (Other)
Responsible Party: Sponsor-Investigator, Yuanjun Yang, director, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CKDRIC-01
Record Dates: First submitted 2024-06-16; First posted 2024-07-15 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases
Keywords: remote ischemic conditioning; chronic kidney disease; renal function
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): The RIC protocol involves five cycles of alternating inflation of both upper arms, utilizing an automated device to alternately inflate to 200 mmHg for 5 minutes and deflate for 5 minutes.
  Interventions: Device: Remote ischemic conditioning
- sham-RIC group (Sham Comparator): The sham-RIC protocol involves five cycles of alternating inflation of both upper arms, utilizing an automated device to alternately inflate to 60 mmHg for 5 minutes and deflate for 5 minutes.
  Interventions: Device: Remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning — RIC is a non-invasive therapy that performed by an electric auto-control device with cuff placed on arm. RIC procedure during which bilateral arm cuffs are inflated to a pressure of 200mmHg for five cycles of 5 min followed by 5 min of relaxation of the cuffs.

SUMMARY:
The incidence of Chronic kidney disease (CKD) is showing an upward trend, but the therapeutic effect of treatment is limited. Remote ischemic conditioning (RIC) has the potential to safeguard remote organs via the repeated application of brief ischemic stimuli. the aim of our study is to investigate whether RIC can protect the renal function in patients with CKD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is characterized by progressive and irreversible loss of nephrons. Currently, due to the increasing prevalence of diabetes, hypertension, obesity, and the impact of population aging, the incidence of CKD is showing an upward trend. The treatment of CKD is mostly aimed at delaying the progression of renal function, but the therapeutic effect is limited, causing a continuous economic burden for CKD patients. Therefore, there is an urgent need to develop new treatment methods to prevent or reverse the progression of the disease.

Remote ischemic conditioning (RIC) is a process that involves repeatedly applying brief ischemic stimuli to a certain organ or tissue, which stimulates the body's endogenous anti-ischemic injury ability, enabling other organs or tissues besides the stimulated one to adapt to ischemia and improve their tolerance to ischemic injury, thereby reducing the damage caused by ischemia to relevant organs or tissues. Current studies have confirmed that RIC can protect remote organs such as the heart, brain, and kidneys through multiple pathways, including humoral mechanisms, neural conduction regulation mechanisms, and immune inflammatory regulation mechanisms. However, current research in the field of kidney diseases has been mostly limited to acute kidney injury caused by contrast agents, surgery, etc., and there are no reports on the intervention and treatment of CKD patients using RIC. Therefore, exploring whether RIC can delay the progression of renal function in CKD patients is of great significance.

ELIGIBILITY:
Inclusion Criteria:

1. CKD Patients with eGFR ≥ 15ml/min/1.73m2
2. Age ≥ 18 years old
3. 24-hour urine protein excretion ≤ 3.5g
4. Subjects who have signed the informed consent form

Exclusion Criteria:

1. Patients with nephrotic syndrome
2. Patients with acute kidney injury
3. Patients who have undergone renal replacement treatment in the past
4. Patients who may have medication changes during RIC or sham-RIC intervention
5. Patients with a history of diabetes or glycated hemoglobin > 8%
6. Patients with familial hypercholesterolemia (>5.5 mmol/L) accompanied by high low-density lipoprotein (>2.5 mmol/L)
7. Patients with contraindications to RIC, such as vascular injury, soft tissue injury, fracture, infection, or known peripheral vascular disease in both arms
8. Patients with a history of hemostatic disorders, systemic bleeding, or thrombocytopenia
9. Patients with cardiogenic embolism (atrial fibrillation) or other severe arrhythmias (severe bradycardia, third-degree atrioventricular block, or ventricular tachycardia), previous myocardial infarction, or severe heart failure (New York Heart Association Class III and IV)
10. Uncontrolled hypertension (defined as systolic blood pressure ≥ 200 mmHg despite antihypertensive treatment)
11. Patients with respiratory failure, malignant tumors, or other autoimmune diseases
12. Women who are pregnant or breastfeeding at the time of enrollment or any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
change in eGFR | 3 months and 12 months
  eGFR is calculated using the CKD-EPI formula, eGFR in mL/min/1.73m²

SECONDARY OUTCOMES:
Changes in renal tissue oxygen saturation (SrtO2) compared to baseline. | 3 months and 12 months
  SrtO2 is measured by Near Infrared Spectroscopy
Changes in blood pressure | 3 months and 12 months
  blood pressure in mmHg

OTHER OUTCOMES:
24-hour urine protein quantitation compared to baseline. | 3 months and 12 months
  The 24-hour urine protein quantitation is monitored through urine.
change in Pulse Wave Velocity compared to baseline. | 3 months
  brachial-ankle Pulse Wave Velocity in cm/s
change in Flow-mediated vasodilation compared to baseline. | 3 months
  FMD in %

CONTACTS AND LOCATIONS:
Overall Officials: Guangyan Cai, Study Director — Chinese PLA General Hospital
Locations (1):
- chinese PLA general hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Ruiz-Ortega M, Rayego-Mateos S, Lamas S, Ortiz A, Rodrigues-Diez RR. Targeting the progression of chronic kidney disease. Nat Rev Nephrol. 2020 May;16(5):269-288. doi: 10.1038/s41581-019-0248-y. Epub 2020 Feb 14. PMID 32060481
- [Background] Zhou D, Ding J, Ya J, Pan L, Wang Y, Ji X, Meng R. Remote ischemic conditioning: a promising therapeutic intervention for multi-organ protection. Aging (Albany NY). 2018 Aug 16;10(8):1825-1855. doi: 10.18632/aging.101527. PMID 30115811
- [Background] Zhang YN, Dai YJ, Cui Y, Wu Q, Zhang NN, Chen HS. Diabetes, fasting blood glucose and the efficacy of remote ischaemic conditioning: A secondary analysis of the RICAMIS trial. Diabetes Obes Metab. 2023 Sep;25(9):2689-2696. doi: 10.1111/dom.15156. Epub 2023 Jun 8. PMID 37288603